CLINICAL TRIAL: NCT04124536
Title: Z 31901 - Combination Partner HIV Testing Strategies for HIV-positive and HIV-negative Pregnant Women: A Pilot Study
Brief Title: Combination Partner HIV Testing Strategies for HIV-positive and HIV-negative Pregnant Women
Acronym: MP3 Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-0276; R01AI131060 (NIH)
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Results first posted 2021-05-24 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-04

CONDITIONS: HIV
Keywords: Self Testing; Partner notification; Secondary Distribution
MeSH Terms: interventions — Contact Tracing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): In addition to standard partner notification services, the intervention arm will receive HIV self-test kits and structured counseling about HIVST, regardless of HIV status.
  Interventions: Behavioral: HIV self-testing with partner notification.
- Control (No Intervention): Standard partner notification services, regardless of HIV status.

INTERVENTIONS:
Behavioral: HIV self-testing with partner notification. — HIV self-test kits are oral swabs. Partner notification will be offered to all women in the intervention arm, regardless of HIV status.
  Arms: Intervention

SUMMARY:
The overall objective of this study is to evaluate whether the addition of secondary distribution HIV self-test kits to existing partner notification guidelines increases the proportion of male partners who access facility-based HIV testing services, when compared to the partner notification strategy alone

DETAILED DESCRIPTION:
Pregnant women 18 years of age or older who enter antenatal care at Chipata Level 1 Hospital in Lusaka, Zambia will participate.

HIV-positive and HIV-negative pregnant women will be randomized to one of two groups: partner notification alone or partner notification plus secondary distribution of HIV self-test kits. Women will return to the clinic 30 days after enrollment for an exit visit during which time information about their experience with the partner notification strategies will be collected.

A random sample of women and health care workers will also participate in qualitative interviews.

ELIGIBILITY:
Inclusion Criteria

* 18 years of age or older
* Pregnant at time of enrollment based on antenatal record
* Documented HIV status (either positive or negative) in antenatal record
* Reports at least one current sexual partner
* Willingness to provide her own contact information
* Ability and willingness to provide informed consent
* Intent to remain in current geographical area of residence for the duration of follow-up activities
* Willingness to adhere to study procedures

Exclusion Criteria

* Women who express concerns about IPV or social harms as a result of participation during the screening process will not be included.
* Women who have previously enrolled in the study will not be permitted to enroll again.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 341 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2020-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ben Chi, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Chipata Health Centre, Lusaka, Zambia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: 9 to 36 months following publication
Access Criteria: IRB, IEC, or REB approval, as applicable, and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Derived] Mutale W, Freeborn K, Graybill LA, Lusaka MM, Mollan KR, Mweemba O, Kasaro M, Lungu R, Kumwenda A, Saidi F, Powers KA, Maman S, Rosenberg NE, Chi BH. Addition of HIV self-test kits to partner notification services to increase HIV testing of male partners of pregnant women in Zambia: two parallel randomised trials. Lancet Glob Health. 2021 Dec;9(12):e1719-e1729. doi: 10.1016/S2214-109X(21)00393-4. Epub 2021 Nov 1. PMID 34735862

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV-Positive Intervention; HIV-Negative Intervention: Combination strategy for partner HIV testing
  HIV self-testing with partner notification. HIV self-test kits are oral swabs. Partner notification will be offered to all women in the intervention arm.
- HIV-Positive Control: Single strategy for partner HIV testing
  Standard partner notification services.
- HIV-Negative Control: Single strategy for partner HIV testing
  Partner notification services adapted for partners of HIV-negative women.
- Healthcare Workers: Healthcare workers were interviewed about the trial interventions, to gain insights into its feasibility.
Period: Overall Study
Arm/Group | HIV-Positive Intervention | HIV-Positive Control | HIV-Negative Intervention | HIV-Negative Control | Healthcare Workers
Started | 58 | 58 | 105 | 105 | 15
Completed | 47 | 53 | 102 | 98 | 15
Not Completed | 11 | 5 | 3 | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthcare Workers: Healthcare workers who were involved in different aspects of male partner HIV testing and included study staff members.
- Total: Total of all reporting groups
Arm/Group | HIV-Positive Intervention | HIV-Positive Control | HIV-Negative Intervention | HIV-Negative Control | Healthcare Workers | Total
Number analyzed (Participants) | 58 | 58 | 105 | 105 | 15 | 341
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 26 [23 to 30] | 26 [23 to 29] | 24 [21 to 28] | 25 [22 to 28] | 37 [34 to 48] | 25 [22 to 29]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 58 | 105 | 105 | 13 | 339
  Male | 0 | 0 | 0 | 0 | 2 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Zambia | 58 | 58 | 105 | 105 | 15 | 341

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Reported Primary Male Partner Completed HIV Testing at a Healthcare Facility
Description: The number of participants who report their primary male partners getting tested for HIV at a healthcare facility when presented with partner notification plus secondary distribution of HIV self-test kits compared to partner notification alone
Time Frame: Enrollment - 30 days post enrollment of study participant
Population: Data reported for all participants with a follow-up visit within 90 days of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-Positive Intervention | HIV-Positive Control | HIV-Negative Intervention | HIV-Negative Control
Number analyzed (Participants) | 47 | 53 | 102 | 98
Participants | 3 | 15 | 3 | 33
Statistical Analysis 1: Comparison: HIV-Positive Intervention vs HIV-Positive Control; Test type: Superiority; Risk Difference (RD) = -21.9, 95% CI 2-sided [-35.9 to -7.9] — The risk difference was calculated by subtracting the proportion of women meeting the outcome in the intervention arm minus the proportion of women meeting the outcome in the control arm
Statistical Analysis 2: Comparison: HIV-Negative Intervention vs HIV-Negative Control; Test type: Superiority; Risk Difference (RD) = -30.7, 95% CI 2-sided [-40.6 to -20.8] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Number of Participants Who Reported HIV Testing With Primary Male Partner at a Healthcare Facility
Description: The number of couples getting tested for HIV when presented with partner notification plus secondary distribution of HIV self-test kits will be compared to partner notification alone.
Time Frame: Enrollment - 30 days post enrollment of study participant
Population: Data reported for all participants with a follow-up visit within 90 days of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-Positive Intervention | HIV-Positive Control | HIV-Negative Intervention | HIV-Negative Control
Number analyzed (Participants) | 47 | 53 | 102 | 98
Participants | 1 | 4 | 0 | 9
Statistical Analysis 1: Comparison: HIV-Positive Intervention vs HIV-Positive Control; Test type: Superiority; Risk Difference (RD) = -5.4, 95% CI 2-sided [-13.6 to 2.8] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: HIV-Negative Intervention vs HIV-Negative Control; Test type: Superiority; The calculation of risk differences between study arms was originally planned. However, the linear-binomial model did not converge because of zero events in the intervention arm

3. Secondary Outcome: Number of Participants Reporting Social Harms
Description: The number of participants reporting social harms associated with the HIV testing approaches. Participants were asked about social harms related to trial participation, including perceived stigma, discrimination, and intimate partner violence.
Time Frame: Enrollment - 30 days post enrollment of study participant
Population: Data reported for all participants with a follow-up visit within 90 days of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-Positive Intervention | HIV-Positive Control | HIV-Negative Intervention | HIV-Negative Control
Number analyzed (Participants) | 47 | 53 | 102 | 98
Participants | 0 | 1 | 0 | 0

4. Secondary Outcome: Number of Healthcare Providers Describing Feasibility of Intervention Via In-depth Interviews (Qualitative)
Description: To gain deeper insights about the feasibility of male partner HIV testing strategies, healthcare workers from the study site were asked to participate in in-depth interviews. Participating healthcare workers were involved in different aspects of male partner HIV testing and included study staff members. Feasibility was defined as a positive rating about the intervention's potential performance in real-life conditions at the clinic and community levels.
Time Frame: 6 months after the start of enrollment
Population: Healthcare workers involved in the provision of male partner HIV testing were interviewed to gain insights about the intervention's feasibility.
Measure: Count of Participants; unit: Participants
Groups:
- Healthcare Workers: Healthcare workers who participated in in-depth interviews were involved in different aspects of male partner HIV testing and included study staff members.
Arm/Group | Healthcare Workers
Number analyzed (Participants) | 15
Participants
  Feasibility of partner notification for HIV-positive women | 9
  Feasibility of partner notification for HIV-negative women | 13
  Feasibility of HIV self-testing for HIV-positive women | 10
  Feasibility of HIV self-testing for HIV-negative women | 15

5. Secondary Outcome: Number of Participants Describing Acceptability of Intervention Via In-depth Interviews (Qualitative)
Description: To gain deeper insights about the acceptability of the different male partner HIV testing strategies, subsamples of participants were selected based on study arm (intervention vs. control) and woman's HIV status (positive vs. negative). For the outcome measure, acceptability was defined as a positive rating of male partner HIV testing strategies from participants based on their experiences.
Time Frame: In the first two months of enrollment
Population: This subsample of participants is based on study arm and woman's HIV status.
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-Positive Intervention | HIV-Positive Control | HIV-Negative Intervention | HIV-Negative Control
Number analyzed (Participants) | 11 | 10 | 10 | 8
Participants
  Acceptability of partner notification | 6 | 4 | 5 | 3
  Acceptability of HIV self-testing | 9 | NA — According to the trial design, participants in the control group did not receive HIV self-test kits to distribute to their male partners. As such, they were not in a position to comment on acceptability. | 8 | NA — According to the trial design, participants in the control group did not receive HIV self-test kits to distribute to their male partners. As such, they were not in a position to comment on acceptability.

6. Other Pre Specified Outcome: Number of Participants Who Reported Primary Male Partner HIV Testing Completed at Any Venue
Description: The number of participants who report their primary male partners getting tested for HIV at any venue when presented with partner notification plus secondary distribution of HIV self-test kits (SD-HIVST) compared to partner notification alone
Time Frame: Enrollment - 30 days post enrollment of study participant
Population: Data reported for all participants with a follow-up visit within 90 days of randomization
Measure: Count of Participants; unit: Participants
Arm/Group | HIV-Positive Intervention | HIV-Positive Control | HIV-Negative Intervention | HIV-Negative Control
Number analyzed (Participants) | 47 | 53 | 102 | 98
Participants | 36 | 19 | 80 | 54
Statistical Analysis 1: Comparison: HIV-Positive Intervention vs HIV-Positive Control; Test type: Superiority; Risk Difference (RD) = 40.7, 95% CI 2-sided [23.0 to 58.4] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: HIV-Negative Intervention vs HIV-Negative Control; Test type: Superiority; Risk Difference (RD) = 23.3, 95% CI 2-sided [10.7 to 36.0] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: From study enrollment through follow-up, a total of approximately 30 -90 days.
Description: Adverse events were documented for all pregnant women in the four arms of the primary trial. Because healthcare workers were not recipients of the strategies under evaluation (either in the control or intervention arms), adverse events were not assessed in this group. Instead, healthcare workers underwent interviews to assess the feasibility of these different strategies.
Arm/Group | HIV-Positive Intervention | HIV-Positive Control | HIV-Negative Intervention | HIV-Negative Control
All-Cause Mortality (participants affected / at risk) | 1/58 | 0/58 | 0/105 | 0/105
Serious Adverse Events (participants affected / at risk) | 1/58 | 0/58 | 0/105 | 0/105
Other Adverse Events (participants affected / at risk) | 0/58 | 0/58 | 0/105 | 0/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIV-Positive Intervention (N=58) | HIV-Positive Control (N=58) | HIV-Negative Intervention (N=105) | HIV-Negative Control (N=105)
Maternal death (Infections and infestations) | 1 | 0 | 0 | 0 — Maternal death due to meningoencephalitis due to advanced HIV disease. This condition was deemed unrelated to study participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-17): https://cdn.clinicaltrials.gov/large-docs/36/NCT04124536/Prot_SAP_000.pdf